CLINICAL TRIAL: NCT07231198
Title: Detection of Microplastics in Patients With Periodontitis - a Cross-sectional Study
Brief Title: Detection of Microplastics in Patients With Periodontitis
Acronym: micropl_perio
Status: Not yet recruiting | Type: Observational
Sponsor: Sigmund Freud PrivatUniversitat (Other)
Responsible Party: Principal Investigator, Hady Haririan, Prof., Sigmund Freud PrivatUniversitat
Other Study IDs: 17538733; SFU (Other Grant/Funding Number: SFU)
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Periodontal Diseases; Periodontitis
Keywords: periodontitis; microplastics
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with periodontitis, stage 3 or 4: Status assessment with supragingival cleaning Sample collection with sterile universal curette (steel) from the bottom of the pockets of the 4 deepest gum pockets (ST >= 5mm) pooled in ultrapure water

SUMMARY:
Plastic particles known as microplastics are now a ubiquitous part of the environment. Human exposure to microplastics occurs through the consumption of contaminated food and polluted air, which affect the intestinal system. Several studies have detected the presence of microplastics in various parts of the human digestive system, e.g., in feces. Unfortunately, little is known about the presence of microplastics in the mouth as the primary part of the digestive system. Periodontal pockets can be considered an ideal deposition site for microplastics. Since microplastics are suspected of being an immunomodulatory factor, there is great interest in their presence in subgingival plaque and their possible exacerbation of chronic inflammatory diseases such as periodontitis. The following study aims to clarify the presence, classification, and concentration of microplastics in subgingival plaque. No comparable study has been identified to date.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over
* Gender: Female / male / diverse
* Patients

  * who have been diagnosed with stage III and IV periodontitis.
  * who have not yet started periodontal treatment.
  * who still have at least 20 teeth. Providing written consent to participate in the study.

Exclusion Criteria:

* Patients

  * who have already been treated for periodontitis
  * who have already undergone/begun periodontitis treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with periodontitis, stage 3 or 4, with a full mouth probing score at the Department of Periodontology, Dental Clinics, Sigmund Freud University, Vienna, Austria
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Microplastics | one year
  number of patients with periodontitis with microplastics in periodontal pockets, quantification of microplastic particles in periodontal pockets, qualitative analysis of microplastic

IPD SHARING:
Plan to Share IPD: Yes
microplastic findings

REFERENCES:
- [Background] Ogata Y. Diffusion of the magnetization profile in the XX model. Phys Rev E Stat Nonlin Soft Matter Phys. 2002 Dec;66(6 Pt 2):066123. doi: 10.1103/PhysRevE.66.066123. Epub 2002 Dec 18. PMID 12513363